CLINICAL TRIAL: NCT07314619
Title: Prospective, Multicenter, Single-Arm, Phase Ⅱ Clinical Study on the Efficacy and Safety of Sacituzumab Tirumotecan Combined With Bevacizumab in Platinum-Resistant Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xie Ya, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-NSIP-032
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer (PROC)
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab tirumotecan combined with bevacizumab (Experimental)
  Interventions: Drug: Sacituzumab Tirumotecan Combined with Bevacizumab

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan Combined with Bevacizumab — Sacituzumab Tirumotecan is administered at a dose of 4 mg/kg via intravenous infusion, with a treatment cycle of every 2 weeks, and is given once on Day 1 of each cycle.
  Bevacizumab is administered at a dose of 7.5~15 mg/kg via intravenous infusion, once every 3 weeks.
  Treatment is continued until disease progression or the occurrence of intolerable toxicity.

SUMMARY:
As one of the gynecological malignancies with the highest incidence and mortality rates worldwide, ovarian cancer treatment faces the significant challenge of platinum-resistant recurrence. Patients with platinum-resistant recurrent ovarian cancer (PROC) have an extremely poor prognosis, and the survival benefits of traditional chemotherapy and bevacizumab combination therapy are limited (median progression-free survival [mPFS] is approximately 2-5 months, and 5-year survival rate is 30%-40%). In recent years, the antibody-drug conjugate (ADC) Sacituzumab tirumotecan has shown breakthrough potential. A phase Ⅱ study presented at the 2024 European Society for Medical Oncology (ESMO) Congress demonstrated that for patients with advanced platinum-resistant ovarian cancer (87.5% of whom had platinum resistance) treated with this drug as monotherapy, the objective response rate (ORR) reached 40%, median progression-free survival (mPFS) was 6.0 months, and disease control rate (DCR) was 75%. Furthermore, the ORR increased to 61.5% in patients with high Trop2 expression, and the safety profile was manageable.Based on the preclinical model evidence suggesting that anti-angiogenic drugs can enhance the intratumoral penetration of ADCs, the current study further explores the synergistic effect of Sacituzumab tirumotecan combined with bevacizumab. It aims to improve therapeutic efficacy by optimizing tumor microcirculation and analyze the molecular mechanisms using technologies such as organoids and single-cell sequencing, thereby providing a new strategy to overcome the bottleneck of platinum resistance.

ELIGIBILITY:
Inclusion Criteria:

* 1.Sign a written informed consent form before undergoing any trial-related procedures;
* 2.Female, aged ≥ 18 years;
* 3.Histologically confirmed epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer; with platinum resistance (recurrence within 6 months after the last platinum dose);
* 4.Enrolled subjects must have received at least one but no more than three prior systemic treatment regimens, and the prior regimens may include bevacizumab and/or poly(ADP-ribose) polymerase inhibitors (PARPi);
* 5.For subjects with brain metastases, only those with asymptomatic or symptomatically stable brain metastases are eligible for enrollment;
* 6.ECOG performance status score of 0-1;
* 7.Expected survival time > 6 months;
* 8.Adequate organ function, with subjects required to meet the following laboratory parameters:

  1. Absolute Neutrophil Count (ANC) ≥ 1.5×10⁹/L without the use of granulocyte colony-stimulating factor (G-CSF) within the past 14 days;
  2. Platelet count ≥ 100×10⁹/L without blood transfusion within the past 14 days;
  3. Hemoglobin > 9 g/dL without blood transfusion or use of erythropoietin within the past 14 days;
  4. Total bilirubin ≤ 1.5×Upper Limit of Normal (ULN);
  5. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5×ULN;
  6. Serum creatinine ≤ 1.5×ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 mL/min;
  7. Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5×ULN;
  8. Normal thyroid function, defined as Thyroid-Stimulating Hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects may still be enrolled if their total triiodothyronine (T3) (or free triiodothyronine, FT3) and free thyroxine (FT4) are within the normal range;
  9. Cardiac enzyme profile within the normal range (subjects with isolated laboratory abnormalities deemed clinically insignificant by the investigator may also be enrolled);
* 9.For women of childbearing potential, a negative urine or serum pregnancy test must be obtained within 3 days before the first administration of the study drug (Cycle 1, Day 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women who are not of childbearing potential are defined as those who are postmenopausal for at least 1 year, or have undergone surgical sterilization or hysterectomy;
* 10.For female subjects with fertility potential, they must agree to use effective medical contraceptive measures from the time of signing the informed consent form until 6 months after the last dose of the study drug.

Exclusion Criteria:

* 1.Diagnosis of other malignant diseases within 5 years before the first dose (excluding radically treated basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, and/or carcinoma in situ with radical resection);
* 2.Known presence of active bleeding signs in lesions as shown by endoscopy;
* 3.Currently participating in therapeutic intervention clinical research, or having received other study drugs or treatment with study devices within 4 weeks before the first dose;
* 4.Previous receipt of the following therapies: ADC drugs targeting FR-α, or TROP2-targeted treatments (such as any drug therapy containing topoisomerase I targeting agents, including antibody-drug conjugate (ADC) therapy);
* 5.Systemic treatment with Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion) within 2 weeks before the first dose;
* 6.Occurrence of active autoimmune diseases requiring systemic treatment (e.g., disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years before the first dose. Replacement therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatment;
* 7.Receipt of systemic glucocorticoid therapy (excluding nasal spray, inhaled, or other forms of local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose of the study; Note: Use of physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) is permitted;
* 8.Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* 9.Known hypersensitivity to the drugs used in this study;
* 10.Failure to fully recover from toxicity and/or complications caused by any intervention (i.e., ≤ Grade 1 or return to baseline, excluding fatigue or alopecia) before the start of treatment;
* 11.Known history of human immunodeficiency virus (HIV) infection (i.e., positive HIV 1/2 antibodies);
* 12.Untreated active hepatitis B (defined as positive HBsAg with HBV-DNA copy number exceeding the upper limit of normal of the laboratory in the research center); Note: Hepatitis B subjects meeting the following criteria may also be enrolled: a) HBV viral load < 1000 copies/ml (200 IU/ml) before the first dose, and subjects should receive anti-HBV treatment throughout the study chemotherapy period to prevent viral reactivation; b) For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and negative HBV viral load, prophylactic anti-HBV treatment is not required, but close monitoring for viral reactivation is necessary;
* 13.Subjects with active HCV infection (positive HCV antibodies and HCV-RNA level above the lower limit of detection);
* 14.Receipt of live vaccines within 30 days before the first dose (Cycle 1, Day 1); Note: Receipt of inactivated viral vaccines for seasonal influenza via injection within 30 days before the first dose is permitted; however, intranasal attenuated live influenza vaccines are not allowed;
* 15.Pregnant or lactating women;
* 16.Presence of any severe or uncontrollable systemic diseases, such as:

  1. Significant and severely symptomatic, uncontrollable abnormalities in resting electrocardiogram (ECG) in terms of rhythm, conduction, or morphology, such as complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmia, or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, or chronic heart failure with New York Heart Association (NYHA) classification ≥ Grade 2;
  3. Any arterial thrombosis, embolism, or ischemia (e.g., myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack) occurring within 6 months before enrollment;
  4. Poorly controlled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
  5. History of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose, or current clinically active interstitial lung disease;
  6. Active pulmonary tuberculosis;
  7. Presence of active or uncontrolled infection requiring systemic treatment;
  8. Presence of clinically active diverticulitis, abdominal abscess, or gastrointestinal obstruction;
  9. Liver diseases such as liver cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poorly controlled diabetes mellitus (fasting blood glucose (FBG) > 10 mmol/L);
  11. Urinalysis indicating urine protein ≥ ++, and confirmed 24-hour urine protein quantification > 1.0 g;
  12. Patients with mental disorders who are unable to cooperate with treatment;
* 17.Need for use of strong inhibitors or inducers of cytochrome P450 3A4 enzyme (CYP3A4) within 2 weeks before the first dose and during the study period (use of strong CYP3A4 inhibitors or inducers is not permitted in this study; all subjects must avoid concurrent use of any drugs, herbal supplements, and/or ingestion of such foods known to induce CYP3A4 as much as possible);
* 18.Documented history of severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or corneal disease that impairs delayed corneal wound healing;
* 19.History of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonia requiring steroid treatment, current presence of ILD or non-infectious pneumonia, or suspected ILD or non-infectious pneumonia at screening that cannot be excluded by imaging examination;
* 20.Evidence of medical history, disease, treatment, or abnormal laboratory test results that may interfere with study results, prevent the subject from completing the study, or other circumstances deemed unsuitable for enrollment by the investigator (including other potential risks considered by the investigator that make the subject unfit for participation in this study).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 24 months
  ORR is defined as the percentage of participants with Complete Response or Partial Response per RECIST 1.1 assessed by the investigators.

SECONDARY OUTCOMES:
PFS | Up to 24 months
  PFS is defined as the time from the first administration to the first documented progressive disease (PD) per RECIST 1.1 by investigators or death due to any cause, whichever occurs first.
OS | Up to 24 months
  OS is defined as the time from the first receipt of treatment under the study protocol to the death of the subject due to any reason.
Adverse Events (AEs) | Up to 24 months
  The number of participants experiencing an AE will be assessed

OTHER OUTCOMES:
Correlation between Trop2 expression, TMB level, immune cell subsets, tumor microenvironment, etc. in tumor tissues and therapeutic efficacy | Up to 24 months
  Correlation between Trop2 expression, TMB level, immune cell subsets, tumor microenvironment, etc. in tumor tissues and therapeutic efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China